CLINICAL TRIAL: NCT03244943
Title: Effects of Non-surgical Periodontal Treatment on the Gingival Crevicular Fluid Cytokine Profiles in Breast Cancer Patients Undergoing Chemotherapy
Brief Title: Cytokine Profiles in Breast Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Kelly Rocio Vargas Villafuerte, Master of periodontics, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37030514.7.0000.5419
Record Dates: First submitted 2017-08-04; First posted 2017-08-10 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2017-08

CONDITIONS: Mammary Neoplasm, Human; Periodontal Diseases; Chemotherapy Effect
MeSH Terms: conditions — Breast Neoplasms; Periodontal Diseases | interventions — Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: 40 patients were allocated: periodontitis patients (P) (n=20) and breast cancer with periodontitis patients (CAN/P) (n=20). The clinical parameters: probing depth (PD), clinical attachment level (CAL), plaque index (PI), Bleeding of probing (BOP) and levels of IFN-γ, IL-4, IL-10, TGF-β, IL-17, IL-2, IL-6, IL-1β and TNF-α in gingival crevicular fluid (GCF) were evaluated at baseline, 45 and 180 days after therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non surgical periodontal treatment (Other): The NSPT, which consisted of subgingival debridement - scaling and root planning (SRP) under local anesthesia.
  Interventions: Procedure: Non surgical periodontal Treatment

INTERVENTIONS:
Procedure: Non surgical periodontal Treatment — The NSPT, which consisted of subgingival debridement - scaling and root planning (SRP) under local anesthesia. On average, the treatment of the entire oral cavity was completed within four sessions (sessions of 50 minutes). The SRP was performed by one experienced periodontist (KRVV) using Gracey curettes (Hu-Friedy MFG. Co. Inc., Chicago, IL, USA), ultra-sonic devices (Bob-Cat, Dentsply/Cavitron, Long Island City, NY, USA) and, if necessary, with multilaminated drills.
  Other Names: scaling and root planning (SRP) under local anesthesia.

SUMMARY:
Aim: This study evaluated the effects of non-surgical periodontal therapy (NSPT) on the cytokine profile and the correlation to clinical parameters of patients undergoing chemotherapy for breast cancer.

Materials and methods: 40 patients were allocated: periodontitis patients (P) (n=20) and breast cancer with periodontitis patients (CAN/P) (n=20). The clinical parameters: probing depth (PD), clinical attachment level (CAL), plaque index (PI), Bleeding on probing (BOP) and levels of IFN-γ, IL-4, IL-10, TGF-β, IL-17, IL-2, IL-6, IL-1β and TNF-α in gingival crevicular fluid (GCF) were evaluated at baseline, 45 and 180 days after therapy.

DETAILED DESCRIPTION:
The NSPT, which consisted of subgingival debridement - scaling and root planning (SRP) under local anesthesia. On average, the treatment of the entire oral cavity was completed within four sessions (sessions of 50 minutes). The SRP was performed by one experienced periodontist (KRVV) using Gracey curettes (Hu-Friedy MFG. Co. Inc., Chicago, IL, USA), ultra-sonic devices (Bob-Cat, Dentsply/Cavitron, Long Island City, NY, USA) and, if necessary, with multilaminated drills.

ELIGIBILITY:
Inclusion Criteria:

* All patients were diagnosed with periodontitis (P) The inclusion criteria were:Loss of clinical insertion (CAL) ≥ 5mm and PD probing depth ≥ 6mm in ≥ 30% of sites; ≥20 teeth; radiographic bone loss that extends to the middle level of the root; presence of supragingival and subgingival calculus according to the severity of periodontal damage. Grade B was assessed indirectly, considering radiographic bone loss in the tooth most affected by dentition as a function of age (0.25 to 1.0).

Exclusion Criteria:

* 1) scaling and root planning or antibiotic treatment in the previous 6 months; 2) systemic diseases that could affect the progression of periodontitis (e.g., diabetes, hypertension, cardiovascular diseases); 3) extensive prosthetic involvement; 4) long-term administration of anti-inﬂammatory medication; 6) smokers and former smokers; 7) pregnancy or lactation; 8) orthodontic therapy; 9) use of mouth rinses containing antimicrobials in the preceding 2 months; 10) patients had previously received chemotherapy or radiotherapy; 11) patients with metastasis and/or patients with neoadjuvant chemotherapy.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with cancer and without breast cancer between 35 and 70 years of age
Enrollment: 40 (Actual)
Dates: Start 2015-08-01; Primary Completion 2016-12-12 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Cytokines | baseline, 45 days, 180 days
  Cytokine levels and changes before and after post treatment

SECONDARY OUTCOMES:
Correlation of cytokines | baseline, 45 days, 180 days
  cytokine levels between parameters clinical

IPD SHARING:
Plan to Share IPD: Yes
De- identified individual participant for all primary and secundary outcome measures will be made available
Supporting Information: Study Protocol
Time Frame: 6 months of study completion
Access Criteria: data access request will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement